CLINICAL TRIAL: NCT03396302
Title: Impact of An Exercise and Nutritional Education Based Intervention Through New Technologies on Body Composition and Blood Pressure in Hypertensive People With Overweight and Obesity
Brief Title: Lifestyle On-line Intervention in Patients With Obesity and Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-UCH 2017-18
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Hypertension
Keywords: Exercise; Nutrition; Internet; Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension; Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will receive access to the web-based lifestyle intervention (exercise and nutritional education).
  Interventions: Other: Educational intervention
- Control (No Intervention): The control group will receive Hospital treatment as usual.

INTERVENTIONS:
Other: Educational intervention — The self-applied on-line intervention will comprise a three months behavioural intervention composed by 8 modules seeking to develop gradually achieving the goals of changing eating and physical activity habits.
  Other Names: ICT intervention
  Arms: Experimental

SUMMARY:
This study aims to describe a totally self-applied online program to promote healthy lifestyles (nutritional education and exercise practice) for obese participants with hypertension. Participants will be recruited from users of a hypertension unit of a public hospital and will be randomized into two groups: experimental group and control group (treatment as usual). The experimental program (3 months) will be composed by 8 modules aimed for promoting healthy eating habits and increase physical activity. Assessment will include: body composition (BMI), blood pressure, glucose metabolism variables, and physical activity level (measured with accelerometers).

Design: Randomized Controlled Trial.

DETAILED DESCRIPTION:
Healthy eating and regular exercise play an important role to maintain health while ageing. Nutritional education and exercise practice could be monitored by different means, such as Internet, face to face and/or through exercise diaries. Information and Communication Technologies (ICTs) could be a useful tool to promote health, and could be used to work on barriers, such as low motivation and difficulties to maintain exercise or diet. ICTs also have other important advantages, especially their good cost-benefit relationship and the possibility of increasing the efficiency of interventions, allowing them to reach a wider audience at a lower cost. This study aims to describe a totally self-applied online program to promote healthy lifestyles (nutritional education and exercise practice) for obese participants with hypertension. Participants will be recruited from users of a hypertension unit of a public hospital and will be randomized into two groups: experimental group and control group (treatment as usual). The experimental program (3 months) will be composed by 8 modules aimed for promoting healthy eating habits and increase physical activity. Assessment will include: body composition (BMI), blood pressure, glucose metabolism variables, and physical activity level (measured with accelerometers).

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI= 25-35 kg/m2)
* Hypertension

Exclusion Criteria:

* Not having access to the Internet or lack of information about it.
* Treatment with more than 3 antihypertensive drugs.
* Diabetes Mellitus Diagnosis.
* Meet the criteria of the DSM-IV-TR of a Food Disorder.
* Presenting some type of severe psychiatric disorder.
* Disability that prevents or hinders physical exercise.
* Be receiving some treatment for weight loss in another center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
BMI | At three months
  Body mass index

SECONDARY OUTCOMES:
Blood Pressure (BP) | At three months
  Systolic and diastolic blood pressure
Glucose metabolism | At three months
  Levels of glucose (mg/dL) and insulin (mg/dL)
Physical activity | At three months
  Levels of physical activity (measured with accelerometers)

CONTACTS AND LOCATIONS:
Locations (1):
- JF Lisón, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lison JF, Palomar G, Mensorio MS, Banos RM, Cebolla-Marti A, Botella C, Benavent-Caballer V, Rodilla E. Impact of a Web-Based Exercise and Nutritional Education Intervention in Patients Who Are Obese With Hypertension: Randomized Wait-List Controlled Trial. J Med Internet Res. 2020 Apr 14;22(4):e14196. doi: 10.2196/14196. PMID 32286232